CLINICAL TRIAL: NCT00715897
Title: Hyperbaric Oxygen Therapy Induced Neuroplasticity in Post Stroke Patients Suffering Chronic Neurological Deficiencies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Fany Tusia, medical center, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HBOcva1
Record Dates: First submitted 2008-07-14; First posted 2008-07-15 (Estimated); Last update posted 2011-12-26 (Estimated); Status verified 2011-12

CONDITIONS: Chronic Neurological Deficiency; Stroke
Keywords: chronic neurological deficient due to stroke
MeSH Terms: conditions — Stroke | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Treatment- HBOT (Experimental): HBOT treatment: 8-week, 5 times a week administration of 100% O2 for 90 minutes at a pressure of 2 ATA.
  Interventions: Procedure: Hyperbaric Oxygen Therapy (HBOT)
- control-HBOT (No Intervention): Cross group: Patients in the cross group were evaluated three times-baseline, after 2 months control period of no treatment and after a consequent 2 month of HBOT

INTERVENTIONS:
Procedure: Hyperbaric Oxygen Therapy (HBOT) — 8-week, 5 times a week administration of 100% O2 for 90 minutes at a pressure of 2 ATA.
  Arms: Treatment- HBOT

SUMMARY:
The aim of the current work was to evaluate, for the first time in a prospective randomized study, the effect of HBOT on patients with chronic neurological deficiency due to stroke.

DETAILED DESCRIPTION:
Objective: Evaluate the effect of hyperbaric oxygen therapy (HBOT) on patients with chronic neurological deficiency due to stroke.

Methods: A prospective, randomized, control-crossed over trial including patients who had stroke 6-36 months prior to their inclusion. All patients had at least one motor dysfunction. After their inclusion patients were randomized to treated or cross group. The neurologic functions were evaluated by NIHSS, ADL, life quality and brain SPECT. Patients in the treated group were evaluated twice-at baseline and after HBOT. Patients in the cross group were evaluated three times-baseline, after 2 months control period of no treatment and after a consequent 2 month of HBOT. The following HBOT protocol was practice: 40 daily sessions, 90 minutes each, 100% oxygen at 2ATA, 5 days/week,.

Results: The study included 74 patients (8 were excluded). During the control period, in the cross group, NIHSS and the ADL had not changed, while in the treated group both significantly improved. After the cross-over, when the cross group received HBOT, NIHSS and ADL had significantly improved. Same trend of changes were in life quality. The SPECT correlated with the clinical improvement. The improvements were mostly in territories where there was a noticeable discrepancy between the CT and SPECT.

Interpretation: In this study, for the first time, it was demonstrated that HBOT can induce neuroplasticity in patients with chronic neurologic deficiencies due to stroke. The beneficial effect of the HBOT is mostly in territories where there is a brain SPECT/CT mismatch.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older, who had ischemic stroke and 60 patients who had hemorrhagic stroke 6-18 months prior to their inclusion in the study.

Exclusion Criteria:

* Dynamic neurologic improvement or worsening during the last 4 weeks.
* Had been treated with HBO for any other reason prior to their inclusion.
* Have any other indication for HBOT
* Chest pathology incompatible with pressure changes
* Inner ear disease
* Patients suffering from claustrophobia.
* Inability to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2008-08; Primary Completion 2010-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Neurologic evaluation | 2 and 4 months

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Asaf-Harofeh Medical Center, Ẕerifin
  - Research & Development unit, Asaf-Harofeh Medical Center, Ẕerifin

REFERENCES:
- [Derived] Efrati S, Fishlev G, Bechor Y, Volkov O, Bergan J, Kliakhandler K, Kamiager I, Gal N, Friedman M, Ben-Jacob E, Golan H. Hyperbaric oxygen induces late neuroplasticity in post stroke patients--randomized, prospective trial. PLoS One. 2013;8(1):e53716. doi: 10.1371/journal.pone.0053716. Epub 2013 Jan 15. PMID 23335971